CLINICAL TRIAL: NCT04950153
Title: Intensive Combination Approach to Rollback the Epidemic in Nigerian Adolescents: UH3 Phase
Acronym: iCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Babafemi Taiwo, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iCARE Nigeria UH3; UH3HD096920 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Adolescent HIV Infection

STUDY DESIGN:
Intervention Model Description: Stepped wedge (cluster) randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV Testing Intervention (Other): Combination HIV testing and linkage to care intervention includes social media engagement and peer navigation
  Interventions: Behavioral: Social Media Engagement; Behavioral: Testing Peer Navigation
- HIV Treatment Intervention (Other): Combination HIV treatment outcomes (retention, ART adherence and viral suppression) intervention includes SMS text messaging and peer navigation
  Interventions: Behavioral: Peer navigation; Behavioral: SMS Text messaging

INTERVENTIONS:
Behavioral: Peer navigation — Peer navigators will navigate youth with HIV to provide assistance and support to optimize adherence to antiretroviral treatment (ART)
  Arms: HIV Treatment Intervention
Behavioral: SMS Text messaging — Short Message System (SMS) text messages to remind and encourage youth to adhere to their ART
  Arms: HIV Treatment Intervention
Behavioral: Social Media Engagement — HIV testing outreach using social media platforms to promote HIV testing.
  Arms: HIV Testing Intervention
Behavioral: Testing Peer Navigation — Peer navigators will conduct HIV testing outreach and linkage to care to at-risk youth
  Arms: HIV Testing Intervention

SUMMARY:
Combination interventions with mHealth and Peer Navigation components will be evaluated in a randomized, stepped wedge trial among youth in Ibadan, Lagos, Sagamu, and Jos, Nigeria. Study findings will demonstrate whether or not the combination interventions for HIV testing and linkage to care and for HIV treatment outcomes, which were found to be efficacious in our prior pilot UG3 trial, will remain efficacious if scaled as proposed in this UH3 trial, across multiple sites.

DETAILED DESCRIPTION:
A randomized stepped wedge (cluster) trial will be conducted to investigate two combination interventions (each with mHealth + Peer Navigation components) among youth in Ibadan, Lagos, Sagamu, and Jos, Nigeria. Study 1 (Testing and Linkage to Care) will test a combination intervention that targets HIV testing and linkage to care. Study 2 (Treatment Intervention) will test a combination intervention that targets HIV treatment outcomes (retention, adherence and viral suppression).

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV infection
* Registered in the study clinics or their satellite clinics
* On antiretroviral therapy (ART) for at least 3 months
* Intention to remain a study clinic patient during the study observation and intervention period

Exclusion Criteria:

* Inability to provide informed consent
* Youths who are 15 years old and not emancipated, who do not have parental consent

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 558 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
VIral suppression | Week 48
  Proportion of participants with viral suppression, defined as viral load (plasma HIV-1 RNA) <200 copies/ml

SECONDARY OUTCOMES:
Antiretrovial adherence measured by pharmacy drug pick-up | Week 48
  Pharmacy drug pick-up (90% of days with medication)
Antiretroviral drug concentration | Week 48
  Antiretroviral drug concentration in Dried Blood Spot sufficient for viral suppression
Retention in care | Week 48
  Retention, defined as at least two care (non-study) visits in the prior 24-week period

OTHER OUTCOMES:
HIV testing and seroprevalence among young men across multiple sites | Week 48
  HIV seroprevalence among the tested young men during the intervention period (the number of confirmed HIV cases divided by the total number of tests).
Linkage of newly diagnosed young men to a clinic for ART | 48 weeks
  Percentage of young men who are linked to HIV care within 30 days of an HIV confirmatory test

CONTACTS AND LOCATIONS:
Overall Officials: Babafemi Taiwo, MBBS, Principal Investigator — Northwestern University; Robert Garofalo, MD, Principal Investigator — Ann & Robert Lurie Childrens Hospital of Chicago
Locations (6):
- Nigeria (6):
  - University of Ibadan, Ibadan
  - Jos University Teaching Hospital, Jos
  - Lagos State University Teaching Hospital, Lagos
  - Lagos University Teaching Hospital, Lagos
  - Nigerian Institute of Medical Research (NIMR), Lagos
  - Olabisi Onabanjo University Teaching Hospital, Sagamu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kozhumam A, Singh R, Agbaji O, Adetunji A, Taiwo B, Omigbodun O, Kuti K, David A, Akanmu S, Adekambi F, Akinbami A, Oladeji B, Taiwo B, Kuhns LM, Okonkwor O, Berzins B, Johnson AK, Badru T, Janulis P, Adewumi OM, Cervantes M, Awolude O, Garofalo R, Ahonkhai AA, Hirschhorn LR. Attitudes toward scale-up of an Intensive Combination Approach to Rollback the Epidemic in Nigerian adolescents (iCARE) intervention for youth in Nigeria: results of a mixed methods early-implementation study. Implement Sci Commun. 2025 Jan 8;6(1):6. doi: 10.1186/s43058-024-00671-z. PMID 39780298
- [Derived] Taiwo BO, Kuhns LM, Omigbodun O, Awolude O, Kuti KM, Adetunji A, Berzins B, Janulis P, Akanmu S, Agbaji O, David AN, Akinbami A, Adekambi AF, Johnson AK, Okonkwor O, Oladeji BD, Cervantes M, Adewumi OM, Kapogiannis B, Garofalo R. A randomized stepped wedge trial of an intensive combination approach to roll back the HIV epidemic in Nigerian adolescents: iCARE Nigeria treatment support protocol. PLoS One. 2023 Jul 7;18(7):e0274031. doi: 10.1371/journal.pone.0274031. eCollection 2023. PMID 37418498